CLINICAL TRIAL: NCT01977001
Title: Use of MigraineBoxTM Head and Neck Cooling Bath for Treatment of Primary Headache in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 12-3542
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Primary Headache
Keywords: Primary headache; Headache; MigraineBox
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Headache: Treatment with MigraineBoxTM
  Interventions: Device: MigraineBoxTM

INTERVENTIONS:
Device: MigraineBoxTM

SUMMARY:
MigraineBoxTM is a simple, contoured cooling bath for the head and neck. Effectiveness of MigraineBoxTM will be studied in primary headaches in the emergency department. The user simply reclines his/her head and neck into this device that has contours that support the head and neck. Luke warm water is filled into the MigraineBoxTM before use and then a frozen insert is placed inside. This will gradually cool the water surrounding the patient's head and theoretically provide headache relief.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* Benign headache
* Physician intends to treat headache pain in the ED with either droperidol, prochlorperazine, or a parenteral narcotic

Exclusion Criteria:

* Unable to provide informed consent
* Headache due to trauma, subarachnoid hemorrhage, meningitis, intracerebral bleed, cranial tumor, sinusitis, dental pathology, temporomandibular joint dysfunction, glaucoma, or systemic infection
* Known renal impairment
* Known hepatic impairment
* A history of coronary artery disease, peripheral vascular disease, or cerebrovascular disease
* Perforated ear drum
* Pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at an urban county hospital.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain Level | Baseline, 30 minutes, 60 minutes
  Patients will be asked to complete a 100 mm visual analog scale and a four point Likert scale concerning their pain.

SECONDARY OUTCOMES:
Change from Baseline in Nausea | Baseline, 30 minutes, 60 minutes
  Patients will be asked to complete a 100 mm visual analog scale concerning their level of nausea.

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States